CLINICAL TRIAL: NCT01452646
Title: Risk-adapted, MRD-directed Therapy for Young Adults With Newly Diagnosed Acute Myeloid Leukemia. GIMEMA Protocol AML1310. EudraCT Number 2010-023809-36
Brief Title: Risk-adapted, MRD-directed Therapy for Young Adults With Newly Diagnosed Acute Myeloid Leukemia
Acronym: AML1310
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML1310
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; risk-adapted therapy; MRD-directed therapy; young adults
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRD-directed therapy (Experimental)
  Interventions: Other: Risk-adapted, MRD-directed therapy

INTERVENTIONS:
Other: Risk-adapted, MRD-directed therapy — The general objective of this study is that of setting up a multicentre, risk-adapted study that relies on pre-treatment cytogenetic/genetic features and post-consolidation assessment of MRD to establish the final risk assignment and treatment of younger (≤ 60 years) patients with AML. Aim of this clinical trial is to verify whether the delivery of a post remission therapy whose intensity is risk-driven will improve the outcome in terms of both increased anti-leukemic efficacy and reduced therapy-related toxicity.

SUMMARY:
The purpose of this study is to determine whether a risk-adapted, minimal-residual-disease directed therapy for young adults with newly diagnosed acute myeloid leukemia has positive results in terms of overall survival at 24 months.

DETAILED DESCRIPTION:
The general objective of this study is that of setting up a multicentre, risk-adapted study that relies on pre-treatment cytogenetic/genetic features and post-consolidation assessment of Minimal Residual Disease (MRD) to establish the final risk assignment and treatment of younger (≤ 60 years) patients with Acute Myeloid Leukemia (AML). Aim of this clinical trial is to verify whether the delivery of a post remission therapy whose intensity is risk-driven will improve the outcome in terms of both increased anti-leukemic efficacy and reduced therapy-related toxicity.

All patients will receive induction and consolidation chemotherapy according to the Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) LAM99P protocol. After the first consolidation, patients belonging to the low-risk category (core binding factor positive AML without c-Kit mutations, NPM1 positive FLT3 negative AML) will receive autologous stem cell transplantation, patients with high-risk features (adverse-risk karyotype, FLT3-ITD mutations), will be assigned to allogeneic stem cell transplantation. Patients with FLT3-TKD mutations or c-Kit mutated core binding factor positive AML and those belonging to the intermediate-risk karyotype category will be stratified according to MRD by flow cytometry and will receive risk-adapted treatment (autologous vs. allogeneic stem cell transplantation). All patients who meet the criteria for high-risk definition will be offered the allogeneic transplantation option regardless of the availability of a Human Leukocyte Antigen (HLA) identical sibling. In fact, for those lacking a HLA identical sibling all the other sources of hematopoietic stem cells (matched unrelated donor from international registry, unrelated cord blood, family haploidentical donor) will be considered. Autologous or allogeneic stem cell transplantation will be performed within 3 months from the end of consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent according to ICH/EU/GCP and national/local laws
* Patients aged between 18 and 60 years
* Patients previously untreated for their AML by other chemotherapeutic agents (with the exception of no more than 7 days hydroxyurea (HU)), radiotherapy or more than 7 days corticosteroids
* Unequivocal diagnosis of untreated de novo AML according to WHO diagnostic criteria (at least 20% blasts in the bone marrow), with FAB classification other than M3 (acute promyelocytic leukemia), documented by bone marrow aspiration (or biopsy in case of dry tap) (not supervening after other myeloproliferative disease or myelodysplastic syndromes of more than 6 months duration)
* WHO performance status 0-3
* Adequate renal (serum creatinine < 2 x the institutional Upper Limit of Normal (ULN)) and liver (total serum bilirubin < 2 x ULN; serum ALT and AST ≤ 3 x ULN) function, unless considered due to organ leukemic involvement
* Left Ventricular Ejection Fraction (LVEF) >50%, as determined by echocardiogram
* Absence of severe concomitant neurological or psychiatric diseases and congestive heart failure or active uncontrolled infection
* Absence of any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and the follow-up schedule.

Exclusion Criteria:

* Patients aged less than 18 or more than 60 years
* Patients already treated for their AML by other chemotherapeutic agents (with the exception of no more than 7 days HU), radiotherapy or more than 7 days corticosteroids
* Acute promyelocytic leukaemia
* Blast crisis of chronic myeloid leukaemia
* AML supervening after other myeloproliferative disease
* AML supervening after antecedent myelodysplastic syndromes of more than 6 months duration
* Other progressive malignant diseases. However, secondary AML following previously cured malignancies may be included as well as secondary AML following previous exposure to alkylating agents or radiation for other reason
* Inadequate renal or liver function (metabolic abnormalities > 3 times the normal upper limit)
* Severe heart failure requiring diuretics
* Ejection fraction < 50%
* Uncontrolled infections
* WHO performance status = 4
* Severe concomitant neurological or psychiatric diseases
* Patients who are pregnant or adults of reproductive potential not employing an effective method of birth control. Women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to administration of chemotherapy. Post-menopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 515 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Treatment strategy in terms of Overall Survival (OS) at 24 months. | 24 months from study entry.
  OS is defined as the time interval between the date of study entry and death for any cause; patients still alive will be censored at the time of the last follow-up.

SECONDARY OUTCOMES:
Estimation of Disease Free Survival (DFS) from Complete Response (CR) evaluation. | At 24 months from study entry
  DFS is defined as the time interval between the evaluation of CR -after induction phase- and relapse or death in CR; patients still alive, in first CR, will be censored at the time of the last follow-up.
Estimation of Event Free Survival (EFS) from study entry. | at 24 months from study entry
  EFS is defined as the time interval between the date of study entry dose and failure during induction phase, relapse or death whichever comes first; patients still alive, in first CR, will be censored at the time of the last follow-up.
Rate of patients in CR after induction therapy | At 31 days from study entry if pts are in CR or at 69 days from study entry if pts are in PR after 1 induction cycle
Toxicity according to Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0 | From study entry to study completion (6 months therapy + 18 months follow-up)
Estimation of OS, EFS, DFS and Cumulative Incidence of Relapse (CIR) according to risk groups (Low, Intermediate, High) | At 24 months from study entry
  CIR is calculated from the date of achievement of the CR -after induction phase-, using the cumulative incidence method, considering death in CR as a competing risk. Patients still alive, without relapse, will be censored at the time of the last follow-up.
Estimation of OS, EFS, DFS and CIR according to the Minimal Residual Disease (MRD) level at each evaluation step | At 24 months from study entry
Rate of CR patients and estimation OS, EFS, DFS and CIR according to baseline characteristics such as age, performance status, white blood cell (WBC), morphology, cytogenetic and molecular features. | At 24 months from study entry
Quality of Life evaluation | Before treatment starts, after induction, at one year after baseline evaluation.
  QoL should be measured at three different time points:
  1. At Baseline (before treatment starts).
  2. At the end of Induction phase (after evaluation of response and before start of consolidation therapy for patients in CR or salvage therapy for patients not achieving a CR).
  3. At one year after baseline evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Adriano VENDITTI, Pr., Principal Investigator — Policlinico Tor Vergata di Roma
Locations (61):
- Italy (61):
  - U.O. di Ematologia - Azienda Ospedaliera - Pia Fondazione di Culto e di Religione Card. G.Panico, Tricase, (LE)
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma, (RM)
  - Policlinico di Tor Vergata, Rome, (RM)
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - Az. Ospedaliera S. G. Moscati, Avellino
  - Unità Operativa Ematologia 1 - Università degli Studi di Bari, Bari
  - UOC Ematologia Ospedale " Monsignor Raffaele Dimiccoli", Barletta
  - Ist.Ematologia e Oncologia Medica L.e A. Seragnoli, Bologna
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - Servizio di Ematologia - CTMO - ASL 8 P.O. Binaghi, Cagliari
  - Unità Operativa Complessa di Onco-Ematologia - A.O. S.Anna e S.Sebastiano, Caserta
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - Marche U.O. di Medicina Interna - ASUR Marche 8 - Ospedale Civile, Civitanova Alta
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Cona
  - Sezione di Ematologia C.T.M.O. Istituti Ospitalieri, Cremona
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - Clinica Ematologica - Università degli Studi, Genova
  - Divisione di Ematologia Ospedale "Santa Maria Goretti", Latina
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematol, Lecce
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - Ospedale Niguarda " Ca Granda", Milan
  - UO Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Pr. Alfonso Maria D'Arco, Nocera Inferiore
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Ospedale S. Luigi Gonzaga, Orbassano
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - Ospedale Riuniti "Villa-Sofia-Cervello", Palermo
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della MIsericordia, Perugia
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - Azienda ASL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Università di Pisa - Azienda Ospedaliera Pisana - Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Divisione di Ematologia, Pisa
  - Ematologia - Ospedale San Carlo, Potenza
  - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Ospedale S. Camillo, Rome
  - U.O.C. Ematologia - Ospedale S.Eugenio, Rome
  - Sezione di Ematologia Cancer Center Humanitas, Rozzano
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Serv. di Ematologia Ist. di Ematologia ed Endocrinologia, Sassari
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - UOC di Ematologia Generale P.O. S.Vincenzo, Taormina
  - U.O.C. di Ematolgia - A.O. " SS Annunziata" - P.O. S.G. Moscati, Taranto
  - Azienda U.L.S.S.9 - U.O. di Ematologia, Treviso
  - Policlinico Universitario - Clinica Ematologia, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buccisano F, Palmieri R, Piciocchi A, Arena V, Candoni A, Melillo L, Calafiore V, Cairoli R, de Fabritiis P, Storti G, Salutari P, Lanza F, Martinelli G, Luppi M, Capria S, Maurillo L, Del Principe MI, Paterno G, Irno Consalvo MA, Ottone T, Lavorgna S, Voso MT, Fazi P, Vignetti M, Arcese W, Venditti A. ELN2017 risk stratification improves outcome prediction when applied to the prospective GIMEMA AML1310 protocol. Blood Adv. 2022 Apr 26;6(8):2510-2516. doi: 10.1182/bloodadvances.2021005717. PMID 34731884
- [Derived] Venditti A, Piciocchi A, Candoni A, Melillo L, Calafiore V, Cairoli R, de Fabritiis P, Storti G, Salutari P, Lanza F, Martinelli G, Luppi M, Mazza P, Martelli MP, Cuneo A, Albano F, Fabbiano F, Tafuri A, Chierichini A, Tieghi A, Fracchiolla NS, Capelli D, Foa R, Alati C, La Sala E, Fazi P, Vignetti M, Maurillo L, Buccisano F, Del Principe MI, Irno-Consalvo M, Ottone T, Lavorgna S, Voso MT, Lo-Coco F, Arcese W, Amadori S. GIMEMA AML1310 trial of risk-adapted, MRD-directed therapy for young adults with newly diagnosed acute myeloid leukemia. Blood. 2019 Sep 19;134(12):935-945. doi: 10.1182/blood.2018886960. Epub 2019 Aug 8. PMID 31395600
- See also: GIMEMA Foundation Website — http://www.gimema.it/en/index.php